CLINICAL TRIAL: NCT05114759
Title: A Phase I, Open-Label, Multicenter Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of SHR-A2009 for Injection in Patients With Advanced Solid Tumors
Brief Title: A Phase I Clinical Study of SHR-A2009 for Injection in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A2009-I-101
Record Dates: First submitted 2021-10-20; First posted 2021-11-10 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2021-10

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: Single arm study of SHR-A2009
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-A2009 for Injection will be administrated per dose level in which the patients are assigned. (Experimental)
  Interventions: Drug: SHR-A2009

INTERVENTIONS:
Drug: SHR-A2009 — In dose Escalation:
  SHR-A2009 will be administered intravenously. Six dose levels are preset.
  In dose Expansion:
  2 to 3 dose cohorts will be selected for dose expansion stage.
  In indication Expansion:
  Indications will be selected to evaluate preliminary efficacy.

SUMMARY:
This study is an open-label, multicenter Phase I clinical trial to evaluate the safety, tolerability, pharmacokinetics and efficacy of SHR-A2009 for injection in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed unresectable locally advanced or metastatic solid tumors which is relapsed or refractory to standard treatment, or lack of standard treatment, or standard treatment is not applicable currently;
2. Have at least one measurable tumor lesion per RECIST v1.1 (patients with only non-target lesions are allowed to be enrolled in dose escalation stage);
3. ECOG performance status of 0-1;
4. Life expectancy ≥ 12 weeks;
5. Adequate bone marrow and organ function .
6. Subjects must voluntarily agree to participate in the trial and sign a written informed consent form.

Exclusion Criteria:

1. Patients with symptomatic central nervous system metastases or meningeal metastases;
2. Ongoing or previous anti-tumor therapies within 4 weeks prior to the first dose of study drug;
3. Prior treatment with antibody-drug conjugate (ADC) consisting of topoisomerase I inhibitors;
4. History of serious cardiovascular and cerebrovascular diseases;
5. Severe infection within 4 weeks prior to the first dose;
6. Adverse reactions of previous anti-tumor treatment have not recovered to Grade ≤ 1 per NCI-CTCAE v5.0.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) or maximum administered dose (MAD). | From Day 1 to Day 21
  Incidence and category of dose limiting toxicities (DLTs) during the first 21-day cycle of SHR-A2009 treatment.
Recommended Phase 2 dose (RP2D) | From Day 1 to 90 days after last dose
  RP2D will be determined on the basis of evaluation on MTD/MAD, PK, efficacy data in dose escalation and dose expansion stages.
Incidence and severity of adverse events (AEs)/serious adverse events (SAEs) ([CTCAE] v5.0) | From Day 1 to 90 days after last dose
  Assess safety and tolerability of SHR-A2009 by way of adverse events (CTCAE v5.0).

SECONDARY OUTCOMES:
Tmax of SHR-A2009 | approximately 6 months
  Time to maximum concentration of SHR-A2009
Cmax of SHR-A2009 | approximately 6 months
  Maximum concentration of SHR-A2009
AUC0-t of SHR-A2009 | approximately 6 months
  area under the concentration-time curve from time 0 to the last measurable concentration time point of SHR-A2009
AUC0-∞ of SHR-A2009 | approximately 6 months
  area under the concentration-time curve from time 0 to infinity of SHR-A2009
Immunogenicity of SHR-A2009 | approximately 9 months
  Anti-SHR-A2009 antibody (ADA)
Overall response rate (ORR) | approximately within 36 months
  Evaluated using RECIST 1.1
Duration of response (DoR) | approximately within 36 months
  Evaluated using RECIST 1.1
Disease control rate (DCR) | approximately within 36 months
  Evaluated using RECIST 1.1
Progression-free survival (PFS) | approximately within 36 months
  Evaluated using RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (16):
- China (11):
  - Chongqing Cancer Hospital, Chongqicun, Chongqi
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of JiLin University, Changchun, Jlin
  - Shandong Cancer Hospital&Institute, Jinan, Shandong
  - The Second Affiliated Hospital of Air Force Military University Tangdu Hospital, Xi’an, Shanxi
  - Sichuan Cancer Hospital & Institute, Chengdu, Sichuan
  - West China Hospital,Sichuan University, Chengdu, Sichuan
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
- Japan (2):
  - National Cancer Center Hospital East, Chiba
  - National Cancer Center Hospital, Tokyo
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Undecided